CLINICAL TRIAL: NCT07007091
Title: A Phase 1 Pharmacokinetic Study in Healthy Subjects to Evaluate the Bioavailability of Risankizumab Subcutaneous Administration With On-Body Injector Relative to Prefilled Syringe
Brief Title: A Study to Assess the Relative Bioavailability of Risankizumab Following Subcutaneous Administrations With a Pre-Filled Syringe or an On-Body Injector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M25-814
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Risankizumab Prefilled Syringe (PFS) (Experimental): Participants will receive a Subcutaneous (SC) single dose of Risankizumab PFS on Day 1
  Interventions: Drug: Risankizumab
- Arm 2: Risankizumab On-Body Injector (OBI) (Experimental): Participants will receive a Subcutaneous (SC) single dose of Risankizumab OBI on Day 1
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous (SC) Injection
  Arms: Arm 1: Risankizumab Prefilled Syringe (PFS)
Drug: Risankizumab — On-Body Injector (OBI)
  Arms: Arm 2: Risankizumab On-Body Injector (OBI)

SUMMARY:
This study will assess the pharmacokinetics and relative Bioavailability of risankizumab following subcutaneous administration with an on-body injector relative to a prefilled syringe

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is ≥ 18.0 to ≤ 32 kg/m2 after rounding to the tenths decimal at screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Body weight between 40 kg and 100 kg, inclusive, at the time of screening.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* Previous exposure to any anti-interleukin (IL)-12/23 or anti IL-23 treatment for at least one year prior to screening.
* Intention to perform strenuous exercise within one week prior to administration of study treatment and during the study confinement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Risankizumab | Up to Approximately 113 days
  Maximum observed plasma concentration (Cmax) of Risankizumab
Time to Cmax (Tmax) of Risankizumab | Up to Approximately 113 days
  Tmax of Risankizumab
Apparent Terminal Phase Elimination Rate Constant (β) of Risankizumab | Up to Approximately 113 days
  Apparent terminal phase elimination rate constant (β) of Risankizumab
Terminal Phase Elimination Half-life (t1/2) of Risankizumab | Up to Approximately 113 days
  Terminal phase elimination half-life (t1/2) of Risankizumab
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Last Measurable Concentration (AUCt) of Risankizumab | Up to Approximately 113 days
  AUCt of Risankizumab
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Infinity (AUCinf) of Risankizumab | Up to Approximately 113 days
  AUCinf of Risankizumab
Number of Anti-drug antibodies (ADA) | Up to Approximately 113 days
  Incidence of anti-drug antibodies
Number of Participants Experiencing Adverse Events | Up to Approximately 113 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - Cpmi /Id# 276490, Miami, Florida
  - Acpru /Id# 276043, Grayslake, Illinois
  - Ppd - Las Vegas Research Unit /ID# 276565, Las Vegas, Nevada
  - PPD Phase I Clinic /ID# 276525, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-814